CLINICAL TRIAL: NCT00094549
Title: Olanzapine Versus Divalproex and Placebo in the Treatment of Mild to Moderate Mania Associated With Bipolar I Disorder
Brief Title: Olanzapine vs. Comparator and Placebo in the Treatment of Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7029; F1D-MC-HGKQ
Record Dates: First submitted 2004-10-20; First posted 2004-10-21 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Valproic Acid

INTERVENTIONS:
Drug: olanzapine
Drug: divalproex sodium
Drug: placebo

SUMMARY:
The goals of this study are:

A. To determine whether olanzapine can help patients with bipolar disorder who currently have mild to moderate mania.

B. To assess the safety of olanzapine and any side effects that might be associated with it, as well as the quality of life and functioning of patients treated with olanzapine.

C. To assess how olanzapine compares to divalproex.

ELIGIBILITY:
Inclusion Criteria:

* You must be 18 to 65 years old.
* You must have a diagnosis of bipolar I disorder and must be experiencing a manic or mixed (symptoms of mania and depression occurring together) episode.
* You must be able to visit the doctor's office as scheduled for 15 weeks.
* All female patients must test negative for pregnancy and, if of childbearing potential, must be using a medically accepted means of contraception.

Exclusion Criteria:

* You have rapid cycling bipolar disorder, or are having hallucinations or delusions, or are feeling suicidal.
* You are pregnant or breastfeeding
* You have a history of: inadequately controlled diabetes; heart disease; narrow angle glaucoma; low white blood cell or platelet count; have a positive test result for human immunodeficiency virus (HIV+); or any other serious, unstable illnesses as judged by the study physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-10; Study Completion 2006-12

PRIMARY OUTCOMES:
To test the superiority of olanzapine compared with divalproex in improving overall manic symptomatology in patients with mild to moderate
mania associated with bipolar I disorder, as measured by reductions on the Young Mania Rating Scale (YMRS) total score from baseline to the endpoint of Study Period II (3-week acute therapy phase).

SECONDARY OUTCOMES:
Treatment comparison for the reductions of the YMRS total score from baseline to the endpoint of Study Period II: Assess the superiority of olanzapine compared to placebo;
Assess the superiority of divalproex compared to placebo;
In the event that olanzapine vs. divalproex comparison is not significant, and that divalproex is superior to placebo, an assessment of non-inferiority of olanzapine compared with divalproex will be performed
Assess the acute efficacy of olanzapine compared with divalproex and placebo in improving clinical symptomatology during Study Period II, using several measures: Rate of response, with response defined as reduction of
50% or more in the YMRS total score at the endpoint of Study Period II; Time to response, with time to response defined as the time in days from first dose at which a reduction of 50% or more in the YMRS total score is first
observed
given that a response is achieved at the endpoint of Study Period II;
Rate of remission of mania, with remission defined as a YMRS total score of less than or equal to 12 at endpoint of Study Period II; Time to remission of mania, with time to remission defined as the time in days from first
dose at which a YMRS total score of less than or equal to 12 is first observed given that remission is achieved at the endpoint of Study Period II; Reductions from baseline to endpoint of Study Period II on the
Montgomery-Asberg Depression Rating Scale (MADRS) total score and the Clinical Global Impressions-Bipolar Version Severity of Illness (CGI-BP Severity) score
Assess the longer-term efficacy of olanzapine compared with divalproex during Study Period III, using several measures: Reductions in the YMRS, MADRS, and CGI-BP scores from the endpoint of Study Period II to the
endpoint of Study Period III; Rate of failure to maintain response during Study Period III, as measured by a return to a YMRS total score greater than or equal to 20 AND/OR hospitalization due to deterioration in clinical
symptoms of mania at any Study Period III visit, among patients who had achieved response by the endpoint of Study Period II; Time to failure to maintain response during Study Period III, as measured by the time
in days from the endpoint of Study Period II to a return to a YMRS total score greater than or equal to 20 AND/OR hospitalization due to deterioration in clinical symptoms of mania, among patients who had achieved
response by the endpoint of Study Period II; Rate of relapse of mania, where relapse is defined as achieving a YMRS total score greater than or equal to 15 AND/OR hospitalization due to deterioration in clinical symptoms
of mania, at any Study Period III visit, among patients who had achieved remission at the endpoint of Study Period II; Time to relapse of mania, as measured by the time in days from the endpoint of Study Period II to a
return to a YMRS total score greater than or equal to 15 AND/OR hospitalization due to deterioration in clinical symptoms of mania, among patients who had achieved remission at the endpoint of Study Period II
Assess the Treatment by Subgroup interaction of Manic vs. Mixed, as defined by DSM-IV (as assessed by the Clinician's Version of the Structured Clinical Interview for DSM-IV [SCID-CV]), during both Study Period II and
Study Period III for efficacy variables of YMRS and CGI-BP
Assess the rate of switch to a depressive episode in patients not depressed at baseline (MADRS score less than or equal to 12, with a depressive episode defined as a MADRS score greater than or equal to 16 OR
hospitalization due to deterioration in clinical symptoms of depression
Assess the safety of olanzapine compared with divalproex and placebo during Study Period II, and to assess the safety of olanzapine compared with divalproex during Study Period III; Safety evaluations will include
assessment of treatment-emergent adverse events, vital signs and weight, laboratory evaluations, electrocardiograms (ECGs), and extrapyramidal symptoms as assessed using the Barnes Akathisia Scale (Barnes),
Abnormal Involuntary Movement Scale (AIMS), and Simpson-Angus Scale
Evaluate functional status and health-related quality of life associated with olanzapine compared with divalproex as measured by change from baseline to endpoints of Study Period II and Study Period III in
the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36)total score and subscale total scores
Evaluate the level of health resource utilization and resource utilization costs associated with olanzapine compared with divalproex during Study Periods II and III (up to 12 weeks of therapy) using the
Resource Utilization
Assess the rate of hospitalization of patients on olanzapine compared with patients on divalproex during Study Periods II and III (up to 12 weeks of therapy) using the Hospitalization Inventory
Evaluate psychosocial outcomes associated with olanzapine compared with divalproex as measured by change from baseline to endpoints of Study Period II and Study Period III on the Streamlined Longitudinal
Interview Clinical Evaluation from the Longitudinal Interval Follow-up Evaluation (SLICE/LIFE)

CONTACTS AND LOCATIONS:
Overall Officials: Call1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (42):
- United States (31):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Costa Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Pico Rivera, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Boyton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Eagle, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Joliet, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Virginia Beach, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Charleston, West Virginia
- Lithuania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Klaipėda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Šiauliai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Vilnius
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Ziegzdriu K
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Ponce
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Târgu Mureş
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Lipetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Saint Petersburg

REFERENCES:
- [Derived] Houston JP, Kohler J, Bishop JR, Ellingrod VL, Ostbye KM, Zhao F, Conley RR, Poole Hoffmann V, Fijal BA. Pharmacogenomic associations with weight gain in olanzapine treatment of patients without schizophrenia. J Clin Psychiatry. 2012 Aug;73(8):1077-86. doi: 10.4088/JCP.11m06916. PMID 22967772
- [Derived] Houston J, Dharia S, Bishop JR, Ellingrod VL, Fijal B, Jacobson JG, Hoffmann VP. Association of DRD2 and ANKK1 polymorphisms with prolactin increase in olanzapine-treated women. Psychiatry Res. 2011 May 15;187(1-2):74-9. doi: 10.1016/j.psychres.2010.10.020. Epub 2010 Nov 20. PMID 21095016
- [Derived] Tohen M, Vieta E, Goodwin GM, Sun B, Amsterdam JD, Banov M, Shekhar A, Aaronson ST, Bardenstein L, Grecu-Gabos I, Tochilov V, Prelipceanu D, Oliff HS, Kryzhanovskaya L, Bowden C. Olanzapine versus divalproex versus placebo in the treatment of mild to moderate mania: a randomized, 12-week, double-blind study. J Clin Psychiatry. 2008 Nov;69(11):1776-89. doi: 10.4088/jcp.v69n1113. Epub 2008 Oct 7. PMID 19014751